CLINICAL TRIAL: NCT06947928
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial Of IFx-Hu2.0 As An Adjunctive Therapy To Pembrolizumab In Checkpoint-Inhibitor Naïve Participants With Advanced Or Metastatic Merkel Cell Carcinoma
Brief Title: Placebo-Controlled Trial of IFx-Hu2.0 Followed By Pembrolizumab In Checkpoint Inhibitor Naïve Participants With Advanced Or Metastatic Merkel Cell Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TuHURA Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCC 2021-01
Expanded Access: NCT04853602 (Available)
Record Dates: First submitted 2025-04-14; First posted 2025-04-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Or Metastatic Merkel Cell Carcinoma
Keywords: Merkel Cell Carcinoma; Advanced; Metastatic; MCC; pembrolizumab; Innate Immune Agonist; Skin Cancer
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neoplasm Metastasis; Skin Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Participants randomized to the treatment arm will receive IFx-Hu2.0 (0.1 mg) via intralesional injection in a single lesion once per week for 3 consecutive weeks. Pembrolizumab (200 mg) will be administered intravenously (IV) on Day 1, followed by administration every 3 weeks during the first year of treatment. In the second year, the pembrolizumab dose will be 400 mg every 6 weeks. Pembrolizumab treatment will continue until progressive disease (PD), unacceptable immune-related toxicities, or for a maximum duration of 2 years.
  Interventions: Drug: IFx-Hu2.0; Drug: Pembrolizumab
- Control Arm (Placebo Comparator): Participants randomized to the control arm will receive placebo (0.9% Sodium Chloride Injection, USP) via intralesional injection in a single lesion once per week for 3 consecutive weeks. Pembrolizumab (200 mg) will be administered IV on Day 1, followed by administration every 3 weeks during the first year of treatment. In the second year, the dose will be 400 mg every 6 weeks. Pembrolizumab treatment will continue until PD, unacceptable immune-related toxicities, or for a maximum duration of 2 years.
  Interventions: Drug: Placebo; Drug: Pembrolizumab

INTERVENTIONS:
Drug: IFx-Hu2.0 — Therapeutic Classification:
  • Innate immune agonist
  Route of Administration:
  • Intralesional
  Other Names: pAc/emm55
  Arms: Treatment Arm
Drug: Placebo — Route of Administration:
  • Intralesional
  Arms: Control Arm
Drug: Pembrolizumab — Therapeutic Classification:
  • Immunotherapy (Immune checkpoint inhibitor)
  Route of administration:
  • Intravenous (IV) infusion
  Other Names: KEYTRUDA

SUMMARY:
This Phase 2/3, multicenter, randomized, double-blind, placebo-controlled trial will evaluate the Objective Response Rate (ORR) of IFx-Hu2.0 as an adjunctive therapy to pembrolizumab in adult participants (≥18 years) with advanced or metastatic Merkel Cell Carcinoma. A total of 118 participants will be randomized to receive either IFx-Hu2.0 or placebo via intralesional injection in a single lesion, followed by pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Life expectancy equal to or greater than six months.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status < 2.
4. Must be recurrent and/or unresectable Stage III or Stage IV American Joint Committee on Cancer (AJCC) (8th edition) and have histologically confirmed Merkel cell carcinoma

   1. Must have at least one injectable lesion equal to or greater than 3 mm.
   2. Must have measurable disease as defined by RECIST v1.1.
5. Participants should be CPI naïve i.e., no prior therapy with CPI including but not limited to Pembrolizumab, avelumab, ipilimumab, nivolumab.
6. Tumor tissue from an archival core biopsy or resected site of disease must be provided for biomarker analyses. If archival tissue is not available, then a new biopsy should be performed.
7. Adequate hematological, hepatic, and renal function according to laboratory ranges and medical criteria defined within the study protocol.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with protocol requirements.
2. Participants with known active brain metastases with the exception of treated brain metastases that have imaging proving stability at least 4 weeks prior to the start of study treatment, no new metastases, and not requiring steroids.
3. Participants with recurrent resectable MCC
4. Participants with prior systemic chemotherapy
5. Pregnant or breastfeeding females and females desiring to become pregnant or breastfeed within the timeframe of this study.
6. Active, known, or suspected autoimmune disease. Potential Participants with type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll. Low-grade autoimmune toxicity is NOT an exclusion under this criterion.
7. A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks post-treatment initiation and confirmed on a second response assessment at least 28 days after the initial response assessment
  ORR defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) at 12 weeks and confirmed on a second response assessment at least 28 days after the initial response assessment, in the treatment arm based on BICR assessment according to RECIST v1.1. Confirmed response persisting at the time of response assessment, at approximately 24 weeks will constitute the data utilized for the endpoint analysis.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 5 years
  PFS is defined as the time (months) from the date of randomization to the date of the documented PD based on BICR assessment according to RECIST v1.1, or death, whichever occurs first. Participants without progression or death will be censored on the date of last disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Brohl, MD, Principal Investigator — Collaborator
Locations (8):
- United States (8):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Health Care - Skin Cancer Program, Palo Alto, California
  - University of California San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Atlantic Health System, Morristown, New Jersey
  - East Carolina University, Greenville, North Carolina
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington